CLINICAL TRIAL: NCT02714348
Title: Impact of Helminth Infections During Pregnancy on Humoral Vaccine Immunogenicity in Infants
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Centre de Recherche Médicale de Lambaréné (Other)
Collaborators: University Hospital Tuebingen (Other)
Responsible Party: Principal Investigator, Meral Esen, Groupleader immunology and clinical trials, Centre de Recherche Médicale de Lambaréné
Other Study IDs: HelmVacc_II
Record Dates: First submitted 2016-03-16; First posted 2016-03-21 (Estimated); Last update posted 2016-03-21 (Estimated); Status verified 2016-03

CONDITIONS: Maternal Infection Affecting Newborn
Keywords: Helminth infection; Vaccination
MeSH Terms: conditions — Trematode Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Other: Effect of helminth infection on vaccine immunogenicity — Observational; immunology

SUMMARY:
Helminth infection is associated with low vaccine immunogenicity. Pregnant women are particularly sensitive to helminth infection.

Since most vaccines are given shortly after birth, an effect of parasites on infant immunogenicity is of particular concern. Therefore, within this study the investigators aim to investigate if maternal infection influences vaccine immunogenicity in the newborn.

DETAILED DESCRIPTION:
There is evidence that helminth infections during pregnancy affect the immune system of the mother and the unborn child. As a consequence, the antimicrobial- immune and vaccine- response of the infant may be deficient. The aim of the present study is to measure the influence of maternal helminth infection (schistosomal, filarial and intestinal helminth infection) on vaccine immunogenicity of their infants. The main focus is on immune responses of infants to vaccine antigens given as part of the expanded program on immunization (EPI) in Gabon at an age when infants are unlikely to be infected with helminths and are immunologically primed by their intrauterine life. The objective is to investigate if and which species of helminths during pregnancy have an effect on any of the EPI vaccine-induced immune responses.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form (ICF) by the participant aged 18 years or older or by a legal major representative and the participant
* Willingness to deliver in one of the two maternities in the study area
* Willingness and ability to comply with study protocol for the duration of the trial
* Willingness to give blood for the examinations and to provide samples for helminth assessment (stool, urine, blood)

Exclusion Criteria:

* Known chronic diseases (diabetes, TB, HIV, HCV or HBV infection); these will be assessed on a regular basis at given examinations during pregnancy
* Withdrawal of consent
* Poor general health (including a hemoglobin level out of local reference range)
* Signs of symptoms of helminth infection which needs immediate treatment of the mother
* Planned migration from the area

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pregnant women and their infants from Lambaréné and surroundings (Gabon)
Sampling Method: Non-Probability Sample
Enrollment: 323 (Estimated)
Dates: Start 2014-02; Primary Completion 2016-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Difference in Immunoglobulin G (IgG) concentration against EPI vaccine Ags of infants born to helminth infected mothers and non infected mothers at the age of nine months and 12 months | 12 months of observation

CONTACTS AND LOCATIONS:
Overall Officials: Akim A Adegnika, Md, PhD, Study Director — Centre de Recherche Médicale de Lambaréné

IPD SHARING:
Plan to Share IPD: Yes
Publication